CLINICAL TRIAL: NCT01112904
Title: n-3 Fatty Acids and Early Child Nutrition: 5-Year-Olds Follow-Up Study
Brief Title: Essential Fatty Acid (EFA) Nutrition 5-Year-Olds Follow-Up Study
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: H09-01633
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Docosahexanoic Acid (DHA) Status
Keywords: essential fatty acids; DHA status; preschool children; gestation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and blood cells
Oversight: Data Monitoring Committee: No

SUMMARY:
Docosahexanoic acid (DHA) is concentrated in the human brain. Before birth, DHA is transferred across the placenta, but transfer depends on maternal DHA intake. After birth, DHA is provided by breast milk or the child's diet. This study addresses whether DHA intakes are adequate to support human brain development.

In a previous study "N-3 Fatty Acid Requirements for Human Development" (C03-0242), pregnant women were randomly assigned to 400 mg/day DHA or placebo from 16 weeks of gestation until infant delivery. Blood DHA in gestation, and infant development to 18 months were assessed. This follow-up study will assess if maternal DHA in gestation has long-term influence on child development when assessed at 5 years and the impact of the child's own diet.

DETAILED DESCRIPTION:
This research is a prospective follow-up on an existing cohort of women and their children to determine whether dietary intakes of docosahexaenoic acid (DHA) during pregnancy have effects lasting into early childhood. The purpose of this study is to assess the relationship between maternal DHA status in gestation, which is known, and the child 's own diet and relevant genetic variables on the child's neural, cognitive and behavioral development. Hypotheses: 1. maternal DHA status in gestation has a lasting effect on infant development evident when assessed in early childhood 2. Children with low DHA status will be at increased risk for poor scores on tests of development. 3. Genetic variation in fatty acid metabolism will influence blood fatty acids in preschool children.

Objectives: 1. To determine if low maternal DHA status in gestation is related to child development at 5 years of age; 2. To determine the DHA status of children 5 years-of-age in relation to scores on tests of development; 3. To identify the dietary patterns that place children at risk for poor DHA status; 4. To assess if genetic variation in fatty acid metabolism alters blood lipid fatty acids in children This research is a prospective follow-up of 209 children that were last assessed at age 18 months and for whom maternal DHA status in gestation is known. The children with their parents are invited to attend our nutrition lab at the Child and Family Research Institute where the child will complete play-like developmental assessments. Measurement of blood pressure, heart rate, height and weight will be completed and blood samples will be collected to measure DHA, other relevant nutrient that impact development and genetic variables relevant to fatty acids. The parent will provide information on the child' diet and health. Baseline characteristics for the subjects will be summarized using descriptive statistics. Logistic regression will be used to assess the relationship of DHA status to cognitive development with multi-variable-adjusted odds ratios (ORs) of a negative outcome and corresponding 95% confidence interval (CI). Regressions will also be run with the outcomes in continuous form to assess the changes in scores associated with increments of child DHA status. For all multivariate regression models, potential confounders will be screened in stepwise fashion, and any covariate with a regression coefficient P-value < 0.05 (two-sided) will be retained. Variables will include gender, birth weight, gestation length, maternal intelligence quotient (IQ), ethnicity, breast-feeding duration, birth order, and dichotomized variables of child health, eating behavior and martial status. Children will grouped in quintiles of DHA status and descriptive statistics will be used to present intakes of total fat, individual fatty acids. ANOVA will be used to determine if genetic variables influence blood DHA status.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who participated in study (REB # C03-0242 and C&W W03-0084)
* who have already provided written consent for re-contact to participate with their 5 year old child.

Exclusion Criteria:

* Mothers who did not participate in the previous study "N-3 fatty acid requirements for human development"
* Mothers who have not provided written consent for re-contact.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Mothers who participated in study (REB # C03-0242 and C&W W03-0084) and who have already provided written consent for re-contact to participate with their 5 year old child will participate in this follow-up study
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2010-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
maternal DHA status in gestation | 16 & 36 weeks gestation
  red blood cell DHA biochemistries

SECONDARY OUTCOMES:
plasma lutein and Red blood cell DHA | 5 years 8 months to 6 years
  plasma lutein and red blood cell DHA biochemistries

OTHER OUTCOMES:
cognitive development with standardized developmental tests | 5 years 8 months to 6 years
  Assessment with the Kaufman Developmental Assessment Battery

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M. Innis, Dr., Principal Investigator — University of British Columbia; Tim Oberlander, MD, Study Director — University of British Columbia
Locations (1):
- Child & Family Research Institute, Nutrition and Metabolism Research Program, Vancouver, British Columbia, Canada